CLINICAL TRIAL: NCT01843270
Title: Appropriate Laryngeal Mask Airway Size in Patients With Overweight: A Comparison of the Actual Body Weight and Ideal Body Weight
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Yonsei University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Prevention
Other Study IDs: 1-2013-0004
Record Dates: First submitted 2013-04-23; First posted 2013-04-30 (Estimated); Last update posted 2014-09-29 (Estimated); Status verified 2014-01

CONDITIONS: General Anesthesia
Keywords: general anesthesia; body weight; laryngeal mask airway size
MeSH Terms: conditions — Body Weight

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- ideal body weight (Experimental): LMA size based on ideal body weight
  Interventions: Device: ideal body weight based size
- actual body weight (Experimental): LMA size according to actual body weight
  Interventions: Device: actual body weight based size

INTERVENTIONS:
Device: actual body weight based size — According randomized allocated group, the laryngeal mask airway is inserted based on actual or ideal body weight-based sizes before the surgery.
  Arms: actual body weight
Device: ideal body weight based size — According randomized allocated group, the laryngeal mask airway is inserted based on actual or ideal body weight-based sizes before the surgery.
  Arms: ideal body weight

SUMMARY:
The classic laryngeal mask airway is one of the keystones of modern anaesthetic practice. It achieves a reliable airway with a low incidence of major complications and pharynges-laryngeal morbidity. The manufactures of laryngeal mask airway recommend the proper size selection by actual body weight. It was recommended a size 3 for 30-70kg, a size 4 for 70-90 kg, and size 5 for > 90 kg. Obesity increases the fat tissue around an upper airway and decreases the pharyngeal cross sectional area. Also it was reported that pharyngeal area was reduced according to the increasing of BMI. Therefore, the aim of this study is to determine which of actual body weight or ideal body weight is proper on the size selection of laryngeal mask airway.

ELIGIBILITY:
Inclusion Criteria:

* age 20~70
* body mass index > 25 kg/m2
* patient who needs surgery with laryngeal mask airway

Exclusion Criteria:

* difficult airway
* upper airway infection or disease of airway
* history of gastroesophageal reflux
* history of head and neck surgery

Ages: 20 Years to 70 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2013-11; Primary Completion 2014-09 (Actual); Study Completion 2014-09 (Actual)

PRIMARY OUTCOMES:
Oropharyngeal leak pressure | 10mins
  Oropharyngeal leak pressure is measured when the airway pressure becomes the plateau state in condition of gas flow 3 L/min and flow out valve 30 cmH2O.

CONTACTS AND LOCATIONS:
Locations (1):
- Severance Hospital, Seoul, Seoul, South Korea

REFERENCES:
- [Derived] Kim MS, Lee JS, Nam SB, Kang HJ, Kim JE. Randomized Comparison of Actual and Ideal Body Weight for Size Selection of the Laryngeal Mask Airway Classic in Overweight Patients. J Korean Med Sci. 2015 Aug;30(8):1197-202. doi: 10.3346/jkms.2015.30.8.1197. Epub 2015 Jul 15. PMID 26240500